CLINICAL TRIAL: NCT04486456
Title: Epidemiological Study on Anemia and Iron Deficiency in Pregnancy in Medical Institutions in Some Areas of China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Huixia Yang, Principle investigator, Peking University First Hospital
Other Study IDs: ERIC STUDY
Record Dates: First submitted 2020-06-16; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Prevalence
Keywords: Iron deficiency; Anemia during pregnancy
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to describe the prevalence of anemia and iron deficiency in pregnancy through a multi-center, prospective follow-up study . To explore the influence factors of anemia and iron deficiency in pregnancy; to explore the influence of anemia and iron deficiency in pregnancy on maternal and fetal outcomes.

DETAILED DESCRIPTION:
1. To understand the epidemiological characteristics of anemia and iron deficiency in pregnancy and describe the epidemiological situation of anemia and iron deficiency.
2. To explore the influence factors of anemia and iron deficiency in pregnancy.
3. To explore the influence of anemia and iron deficiency during pregnancy on the pregnancy outcome of mothers and infants.

ELIGIBILITY:
Inclusion Criteria:

* Regular prenatal check-ups were conducted in the hospitals participating in the study, and pregnant women who planned to give birth in hospital were established a maternity health manual
* 18 years and older
* Patients have to agree to participate by signing a consent

Exclusion Criteria:

* have severe chronic diseases with Pre-pregnancy
* Suffer from severe mental illness

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnancy patients
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Hb | Completed by observation，an average of 1 year
  Proportion of patients with Hb<110g/L

SECONDARY OUTCOMES:
SF | Completed by observation，an average of 1 year
  Proportion of patients with SF<20μg/L

CONTACTS AND LOCATIONS:
Overall Officials: Xia H Yang, Principal Investigator — The First Affiliated Hospital of Peking University

IPD SHARING:
Plan to Share IPD: Undecided